CLINICAL TRIAL: NCT01281462
Title: A Phase 2, Multicenter, Randomized, Double-blind, Comparative Study to Evaluate the Efficacy and Safety of Intravenous Coadministered Ceftaroline Fosamil and NXL104 Versus Intravenous Doripenem in Adult Subjects With Complicated Urinary Tract Infection
Brief Title: Comparative Study of Coadministered Ceftaroline Fosamil and NXL104 vs. Intravenous Doripenem in Adult Subjects With Complicated Urinary Tract Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CXL-MD-02
Record Dates: First submitted 2011-01-13; First posted 2011-01-24 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Urinary Tract Infections
Keywords: complicated Urinary Tract Infection; Acute Pyelonephritis
MeSH Terms: conditions — Urinary Tract Infections | interventions — Ceftaroline; avibactam; Doripenem; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ceftaroline fosamil and NXL104 (q8h) (Experimental)
  Interventions: Drug: Ceftaroline fosamil and NXL104 (q8h); Drug: Placebo
- Ceftaroline fosamil and NXL104 (q12h) (Experimental)
  Interventions: Drug: Ceftaroline fosamil and NXL104 (q12h); Drug: Placebo
- Doripenem (Active Comparator)
  Interventions: Drug: Doripenem; Drug: Placebo

INTERVENTIONS:
Drug: Ceftaroline fosamil and NXL104 (q8h) — 600 mg ceftaroline fosamil/600 mg NXL104 IV coadministered every 8 hours (q8h);
  Other Names: Ceftaroline fosamil and Avibactam(NXL104) (q8h)
  Arms: Ceftaroline fosamil and NXL104 (q8h)
Drug: Ceftaroline fosamil and NXL104 (q12h) — 600 mg ceftaroline fosamil/600 mg NXL104 IV coadministered every 12 hours (q12h);
  Other Names: Ceftaroline fosamil and Avibactam(NXL104) (q12h)
  Arms: Ceftaroline fosamil and NXL104 (q12h)
Drug: Doripenem — 500 mg doripenem IV q8h;
  Arms: Doripenem
Drug: Placebo — On CXL-MD-02, there were (3) treatment arms (meaning a subject could be randomized to 1 of 3 possible treatment regimens). Each treatment arm contained 1 or 2 placebo doses of IV saline in order to preserve the blind.
  Other Names: placebo (saline)

SUMMARY:
This is a study in adult subjects with complicated urinary tract infection (cUTI) comparing treatment with intravenous (IV) coadministered ceftaroline fosamil and NXL104 versus treatment with IV doripenem.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following inclusion criteria:

* Have pyuria (white blood cells in the urine)
* Clinical signs and/or symptoms of cUTI (including acute pyelonephritis)
* Have a pretreatment baseline urine culture specimen
* The subject's infection would require initial treatment with IV antibiotics
* The subject must require initial hospitalization to manage the cUTI by the standard of care.

Exclusion Criteria:

Subjects must NOT meet any of the following exclusion criteria:

* History of any hypersensitivity or allergic reaction to any β-lactam (eg, cephalosporins, penicillins, carbapenems)
* Confirmed fungal urinary tract infection
* Intractable UTI anticipated to require more than 10 days of study drug therapy
* Complete, permanent obstruction of the urinary tract\
* Permanent indwelling bladder catheter or instrumentation (including nephrostomy) or current urinary catheter that will not be removed during IV study drug administration
* Suspected or confirmed perinephric or intrarenal abscess
* Suspected or confirmed prostatitis
* Ileal loops or vesico-ureteral reflux
* Impairment of renal function including a calculated CrCl of < 30 mL/min, requirement for peritoneal dialysis, hemodialysis or hemofiltration, or oliguria
* Renal transplantation
* Life expectancy less than 3 months
* Evidence of significant hepatic, hematological, or immunologic disease or dysfunction
* Past or current history of epilepsy or seizure disorder
* Women who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2010-12; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Microbiological response of Microbiologically Evaluable (ME) at Test of Cure (TOC) | 5 to 11 days after last dose of study drug
  The number and percentage of subjects in each treatment group recorded as having a favorable microbiological response in the ME Population at Test-of-Cure (TOC)
Evaluate safety | from administration of first dose of study drug to the Late -Follow -Up (LFU) visit (28 to 42 days after administration of the last dose of study drug)
  Evaluate the safety of coadministered IV ceftaroline fosamil and NXL104 in subjects with cUTI. Summaries of AEs, SAEs, deaths, laboratory evaluations (hematology and coagulation studies, comprehensive metabolic panel, and urinalysis), vital signs, ECGs, and physical examinations will be provided for each treatment group.

SECONDARY OUTCOMES:
Clinical response in CE at Test of Cure | 5 to 11 days after last dose of study drug
  The number and percentage of subjects in each treatment group classified as clinical cure Clinically Evaluable (CE) Population at TOC

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Forest Laboratories
Locations (35):
- United States (5):
  - Investigational Site, La Mesa, California
  - Investigational Site, San Diego, California
  - Investigational Site, Pensacola, Florida
  - Investigational Site, Baltimore, Maryland
  - Investigational Site, Detroit, Michigan
- Bulgaria (4):
  - Investigational Site, Plovdiv
  - Investigational Site, Rousse
  - Investigational Site, Sofia
  - Investigational Site, Varna
- Germany (8):
  - Investigational Site, Berlin
  - Investigational Site, Freiburg im Breisgau
  - Investigational Site, Giessen
  - Investigational Site, Kassel
  - Investigational Site, Minden
  - Investigational Site, Müllheim
  - Investigational Site, Paderborn
  - Investigational Site, Planegg
- Investigational Site, Beirut, Lebanon
- Poland (10):
  - Investigational Site, Bialystok
  - Investigational Site, Bielsko-Biala
  - Investigational Site, Częstochowa
  - Investigational Site, Katowice
  - Investigational Site, Lodz
  - Investigational Site, Tychy
  - Investigational Site, Warsaw
  - Investigational Site, Wołomin
  - Investigational Site, Wroclaw
  - Investigational Site, Zamość
- Russia (4):
  - Investigational Site, Moscow
  - Investigational Site, Rostov-on-Don
  - Investigational Site, Saint Petersburg
  - Investigational Site, Smolensk
- Turkey (Türkiye) (3):
  - Investigational Site, Diyarbakır
  - Investigational Site, Eskişehir
  - Investigational Site, Izmir